CLINICAL TRIAL: NCT06323629
Title: Recursive Self-feedback Procedures for Improving Spontaneous Speech Production in Patients With Chronic Aphasia
Brief Title: Effects of Recursive Self-feedback on Speech Production in Aphasia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Center for Smart Use of Technologies to Assess Real-world Outcomes (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY006201
Record Dates: First submitted 2024-02-21; First posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Aphasia; Stroke
MeSH Terms: conditions — Aphasia; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adaptive recursive self-feedback procedure (Experimental): Using a tablet, participants listen to speech playback of their response to a prompt and self-correct/minimize their speech errors in a subsequent attempt. This process is looped multiple times per prompt. It adapts across narrative prompts with low and high complexities.
  Interventions: Behavioral: Adaptive recursive self-feedback procedure
- Non-adaptive recursive self-feedback procedure (Experimental): Using a tablet, participants listen to speech playback of their response to a prompt and self-correct/minimize their speech errors in a subsequent attempt. This process is looped multiple times per prompt. However, it only uses narrative prompts with high complexity.
  Interventions: Behavioral: Non-adaptive recursive self-feedback procedure

INTERVENTIONS:
Behavioral: Adaptive recursive self-feedback procedure — The intervention uses self-feedback alone to improve speech production. It adapts the complexity of the treatment tasks.
  Arms: Adaptive recursive self-feedback procedure
Behavioral: Non-adaptive recursive self-feedback procedure — The intervention uses self-feedback alone to improve speech production. However, it does not adapt the complexity of the treatment tasks.
  Arms: Non-adaptive recursive self-feedback procedure

SUMMARY:
The goal of this clinical trial is to test the effects of recursive self-feedback procedures on spontaneous speech production in stroke survivors with impaired speech production (aphasia). The main question it aims to answer is:

• To what extent can stroke survivors with aphasia use their self-feedback alone to improve their spontaneous speech production?

Participants will be engaged in the following activities:

* They will perform language and cognitive tasks.
* Afterwards, they will receive treatments using tablets and headphones at no cost to them.
* The experimental treatments (recursive self-feedback procedures) entails responding to prompts, listening to playbacks of their speech response and attempt to minimize/correct the errors in the next attempt. This process will be repeated multiple times per prompt.
* The experimental treatments are two: an adaptive version that adapts the complexity of the treatment prompt and a non-adaptive version that does not adapt task complexity.
* Researchers will compare the experimental treatments to see if both have similar effects on improving spontaneous speech production.

ELIGIBILITY:
Inclusion Criteria:

* 6 months post left hemisphere stroke
* Aphasia due to left hemisphere stroke
* Dominant English speaker

Exclusion Criteria:

* Speech-language deficits due to neurological insults such as Parkinson's disease, neurodegenerative conditions etc.
* Uncorrected sensory impairments.
* Language comprehension impairment.
* Severe cognitive impairment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Speaking rate | Within 1 week before treatment and within 1 week after treatment.
  Correct words produced per minute
Speech initiation latency in milliseconds | Within 1 week before treatment and within 1 week after treatment.
  Latency before retrieving the first correct word in an utterance.

CONTACTS AND LOCATIONS:
Overall Officials: Gerald C. Imaezue, PhD, Principal Investigator — University of South Florida

IPD SHARING:
Plan to Share IPD: No
Individual participant data will only be shared with approved members of the research team.